CLINICAL TRIAL: NCT05165225
Title: Phase II Neoadjuvant Pyrotinib Combined with Neoadjuvant Chemotherapy in HER2-low-expressing and HR Positive Early or Locally Advanced Breast Cancer: a Single-arm, Non-randomized, Single-center, Open Label Trial
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Chang Gong, Chief physician, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PILHLE-001
Record Dates: First submitted 2021-12-20; First posted 2021-12-21 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer; HER2-low-expressing Breast Cancer; Hormone Receptor-positive Breast Cancer; Neoadjuvant Therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — pyrotinib; Epirubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Pyrotinib (Experimental): Experimental: Patients will receive Pyrotinib combined with Epirubicin and Cyclophosphamide followed by Docetaxel
  Interventions: Drug: Pyrotinib + epirubicin and cyclophosphamide followed by docetaxel treatment

INTERVENTIONS:
Drug: Pyrotinib + epirubicin and cyclophosphamide followed by docetaxel treatment — Drug: Pyrotinib pyrotinib 320mg orally daily Drug: Epirubicin epirubicin 90mg/m^2 d1 iv Q3W for 4 cycles Drug: Cyclophosphamide cyclophosphamide 600mg/m^2 d1 iv Q3W for 4 cycles Drug: Docetaxel docetaxel 100mg/m^2 d1 iv Q3W for 4 cycles

SUMMARY:
This is a single-arm, prospective, non-randomized, single-center, open label clinical study for evaluating the efficacy and safety of neoadjuvant pyrotinib combined with epirubicin and cyclophosphamide followed by docetaxel in HR positive and HER2-low-expressing early or locally advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent for all study according to local regulatory requirements prior to beginning specific protocol procedures
2. Female patients, age ≥ 18 years
3. Histologically confirmed unilateral primary carcinoma of the breast, except for occult breast cancer, inflammatory breast cancer without assessable focus or eczema like breast cancer
4. HER2-low-positive (defined here as HER2 IHC 2+ and FISH-) and HR positive(defined here as ER and/or PR >1% stained cells)
5. Tumour greater than 2 cm diameter or histologically (core- or fine-needle biopsy) involved lymph nodes
6. According to RECIST version 1.1, there is at least one evaluable target lesion
7. Performance Status- Eastern Cooperative Oncology Group (ECOG) 0-1
8. Required laboratory values including following parameters: WBC count:≥3.0 x 10^9/L ; ANC: ≥ 1.5 x 10^9/L; Platelet count: ≥ 100 x 10^9/L; Hemoglobin: ≥ 9.0 g/dL; Total bilirubin: ≤ 1.5 x upper limit of normal (ULN); ALT and AST: ≤ 2.5 x ULN; alkaline phosphatase ≤ 2.5 × ULN; Serum creatinine: ≤ 1.5 × ULN; Left ventricular ejection fraction (LVEF) ≥ 55%
9. For female patients without menopause or surgical sterilization: consent to contraception both during the trial and within 6 months after the last administration of the test drug

Exclusion Criteria:

1. Metastatic disease (Stage IV) or bilateral breast cancer
2. Known history of hypersensitivity to pyrotinib or any of it components
3. According to the judgment of the researcher, other anti-tumor treatments (except for ovarian function inhibitors) are required during neoadjuvant therapy
4. Patients with severe heart disease or discomfort who are expected to be unable to tolerate chemotherapy, including but not limited to these: 1). Fatal arrhythmia or higher grade atrioventricular block (second degree type 2 atrioventricular block or third degree atrioventricular block) 2). Unstable angina pectoris 3). Heart valve disease with clinical significance 4). ECG showed transmural myocardial infarction pain 5). Poor control of hypertension
5. Patients underwent major breast cancer-free surgery within 4 weeks or have not fully recovered
6. Serious or uncontrolled infections that may affect study treatment or evaluation of study results, including but not limited to active hepatitis virus infection, human immunodeficiency virus (HIV) antibody positive, lung infection, etc
7. History of other malignant tumors in the past 5 years (excluding cured carcinoma in situ of cervix or skin basal cell carcinoma)
8. Those with basic gastrointestinal diseases (especially long-term history of diarrhea or/and constipation)；Inability to swallow、intestinal obstruction or other factors will affect drug administration and absorption
9. The investigator believes that the patient has any other conditions that are not suitable for participation in the study

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2021-07-13 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Residual cancer burden 0/1 (RCB-0/1) rate | within 6 weeks after surgery
  The percentage of patients with RCB-0/1 after neoadjuvant therapy

SECONDARY OUTCOMES:
Pathological complete response (pCR) rate | within 6 weeks after surgery
  The percentage of patients with pCR (ypT0/is, ypN0) after neoadjuvant therapy
Objective response rate (ORR) | within 6 weeks after surgery
  The percentage of subjects with CR or PR as the best response during the period from the beginning of the treatment to the progression of the disease or the completion of preoperative neoadjuvant therapy 【(CR+PR)/Analysis of the total number of people】
Breast conservation rate. | within 6 weeks after surgery
  The breast conservation rate after treatment.
Disease-free Survival (DFS) | 5 years
  The DFS is defined as the time from registration until any relapse, secondary malignancy, or death from any cause
Overall Survival (OS). | 5 years
  The OS is defined as the time from registration to death, irrespective of cause.
Biomarkers | 5 years
  Biomarkers: e.g. Tils
Incidence of grade 3-5 diarrhea. | before surgery
  Diarrhea were graded according to the National Cancer Institute's Common Toxicity Criteria for Adverse Events (CTCAE) version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Gong - Chang, doctor, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No